CLINICAL TRIAL: NCT03797521
Title: A Phase 2, Double Blind, Placebo-Controlled Study to Explore the Safety, Tolerability, and Activity of SXC-2023 in Adults With Moderate to Severe Trichotillomania (TTM) When Dosed for 6 Weeks
Brief Title: A Study in Patients With Trichotillomania
Acronym: TTM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Promentis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-201
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Trichotillomania
Keywords: Promentis Pharmaceuticals; TTM; SXC-2023
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Placebo-controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SXC-2023 50mg QD (Experimental): SXC-2023 50mg dosed once daily for 6 weeks
  Interventions: Drug: SXC-2023
- SXC-2023 200mg QD (Experimental): SXC-2023 200mg dosed once daily for 6 weeks
  Interventions: Drug: SXC-2023
- SXC-2023 800mg QD (Experimental): SXC-2023 800mg dosed once daily for 6 weeks
  Interventions: Drug: SXC-2023
- Matching Placebo QD (Placebo Comparator): Matching Placebo dosed once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SXC-2023 — SXC-2023 oral capsules
  Arms: SXC-2023 200mg QD; SXC-2023 50mg QD; SXC-2023 800mg QD
Drug: Placebo — Matching Placebo oral capsules
  Arms: Matching Placebo QD

SUMMARY:
The purpose of this study is to explore the safety, tolerability and activity of SXC-2023 when dosed for 6 weeks versus placebo in adult patients with moderate to severe Trichotillomania.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, double-blind, placebo-controlled, parallel-group study consisting of a screening period of up to 40 days, a 6 week randomized double-blind treatment period, followed by an up to 2 week safety follow-up period after the last dose of study medication.

Patients will be randomized to one of four treatment groups. Patients will participate for a total of up to 10 weeks, including screening, the 6-week treatment period and follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Adult, female or male, 18-45 years of age, inclusive at screening.
2. Provided signed written informed consent with willingness and ability to comply with all aspects of the protocol.
3. Diagnosis of current TTM based on Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria and confirmed using the clinician-administered MINI-TTM. In addition, subjects should:

   1. Have a history of TTM for at least one year
   2. Have a history of daily hair pulling for at least 6 months prior to the first dose
4. Except for SSRIs or SNRIs, has not used any psychoactive medications including, but not limited to, other antidepressants, anxiolytics, mood stabilizers, anti-psychotics, benzodiazepines, stimulants, sulfasalazine, and St. John's Wort 30 days prior to first dose. Subjects will be allowed to maintain background therapy with SSRIs or SNRIs if on stable regimen for a minimum of 90 days prior to first dose and there are no anticipated changes to the SSRI/SNRI during course of trial.
5. Has not used N-acetylcysteine for at least 90 days prior to the first dose.
6. Has not used gemfibrozil or repaglinide for 1 week prior to the first screening visit.
7. Medically healthy with no clinically significant findings in medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the Principal Investigator (PI) or designee.
8. For a female of childbearing potential: either be sexually inactive (abstinent as a life style) for 28 days prior to the first dosing and throughout the study or be using one of the following acceptable birth control options:

   * Oral contraception for at least 3 months prior to the first dosing along with either a physical (e.g., condom, diaphragm) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study
   * IUD (either hormone-releasing or non-hormone releasing) for at least minimum duration per current labeling along with either a physical (e.g., condom, diaphragm) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study
   * Depo contraception for at least minimum duration per current labeling prior to the first dosing along with either a physical (e.g., condom, diaphragm) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study
   * Double physical barrier method (e.g., condom and diaphragm) from 14 days prior to the first dose and throughout the study
   * Physical plus chemical barrier method (e.g., condom with spermicide) from 14 days prior to the first dose and throughout the study.

   In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 30 days following the last dose.
9. Female of non childbearing potential: must have undergone one of the following sterilization procedures, at least 6 months prior to the first dose:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; Or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum follicle stimulating hormone levels consistent with postmenopausal status or have medically documented history of biological or congenital sterility.
10. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 30 days beyond the last dose of study drug/placebo.
11. If male, must agree not to donate sperm from the first dose until 30 days after the last dose administration.
12. Must be able to fluently read and write in English.
13. Understands the study procedures in the informed consent form (ICF) and is willing and able to comply with the protocol.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding or intend to become pregnant during the study period or within 30 days of the final dose of study drug.
2. Subjects engaged in cognitive behavioral therapy (CBT) for TTM or other body-focused repetitive behavior or any obsessive-compulsive related or impulse control disorder any time within 60 days prior to first dose. For other psychotherapies, subject must have been engaged in that psychotherapy for a minimum of 60 days at the time of first dose and must be willing to maintain the same frequency and type of therapy for the duration of the study period.
3. Subjects engaged in any other behavioral interventions (e.g., wearable devices, behavioral self-help strategies) within 60 days prior to first dose.
4. Mentally or legally incompetent.
5. Suffered a concussion in the past 6 months prior to screening. Any history of traumatic brain injury with loss of consciousness in the year prior to first screening visit.
6. Any lifetime history of any psychotic disorder, including schizophrenia or any bipolar or bipolar-related disorder as determined by clinical history or confirmed at screening with the MINI, version 7.0.2.
7. Current major depressive episode confirmed at screening with the MINI, version 7.0.2.
8. Per PI judgment, the presence of any emotional problems or psychiatric disorders that may obscure evaluation of primary TTM or pose a risk to subject safety or stability during the study period. Other emotional problems or diagnoses may include, but are not limited to, other body-focused repetitive behaviors, post-traumatic stress disorder, obsessive-compulsive disorder, panic disorder, compulsive gambling, borderline personality disorder, or antisocial personality disorder.
9. History of any injury, illness, or condition that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
10. Laboratory evidence of renal impairment (e.g. a creatine clearance of < 80)
11. Presence of any substance use disorder or, in the opinion of the PI or designee, problematic substance use (excluding nicotine or caffeine) within the 2 years prior to screening.
12. History of seizure disorder with the exception of subjects who have been off anti-seizure medication and have not had a seizure in the past 5 years.
13. Subjects with any of the following:

    1. Any psychiatric hospitalizations in the past year,
    2. Imminent risk of suicide based on PI's or designee's clinical judgment or psychiatric examination,
    3. Active suicidal ideation in the past 6 months as evidenced by positive endorsement to Item 4 or 5 on the C-SSRS, OR
    4. Any history of suicidal behavior in the past year as evidenced by positive endorsement to any of the suicidal behavior items on the C-SSRS.
14. Has previously participated in any Promentis Phase 1 study.
15. Participation in another interventional clinical study (including CBT or other behavioral intervention) within 30 days prior to the first screening visit. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to the date of initiation of screening in the current study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Explore the incidence of treatment-emergent adverse events in adults with moderate to severe TTM | Up to 7 weeks
  Safety and tolerability assessed using the frequency of subjects with serious adverse events, adverse events leading to discontinuation, and adverse events judged to be related to study medication.

SECONDARY OUTCOMES:
Change from baseline hairpulling frequency and severity through 6 weeks | Up to 7 weeks
  Improvement will be assessed using the different measurement parameters of all scales using scales such as the Massachusetts General Hospital Hairpulling scale (MGH-HPS)
Change from baseline hairpulling frequency and severity through 6 weeks | Up to 7 weeks
  Improvement will be assessed using the different measurement parameters of all scales using scales such as the Clinical Global Impression of Severity and Change (CGI-S/C)
Change from baseline hairpulling frequency and severity through 6 weeks | Up to 7 weeks
  Improvement will be assessed using the different measurement parameters of all scales using scales such as the Patient Global Impression of Status and Change (PGI-S/C)
Change from baseline hairpulling frequency and severity daily through 6 weeks | Up to 7 weeks
  Improvement will be assessed using the different measurement parameters of all scales using scales such as the Trichotillomania Symptom Diary (TSD)
Preliminary psychometric evidence of the Trichotillomania Symptom Diary (TSD) will be assessed | Up to 7 weeks
  The reliability, validity and responsiveness of the newly developed TSD assessment will be assessed at the item level.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Brostowin, Study Director — Promentis Pharmaceuticals
Locations (13):
- United States (13):
  - CNRI- Los Angeles, Pico Rivera, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Behavioral Clinical Research, North Miami, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Univ of Chicago, Chicago, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Insight Clinical Trials, LLC, Shaker Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Carolina Clinical Trials, Inc, Charleston, South Carolina
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03797521/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03797521/SAP_001.pdf